CLINICAL TRIAL: NCT00005309
Title: Prospective Study of HIV Infection in Hemophiliacs
Status: Completed | Type: Observational
Sponsor: Bloodworks (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 3012; R01HL043512 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2016-02

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections; Blood Disease; Hemophilia A; Hepatitis, Viral, Human; Blood Transfusion; Cytomegalovirus Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Hematologic Diseases; Hemophilia A; Hepatitis, Viral, Human; Cytomegalovirus Infections

SUMMARY:
To examine mechanisms of individual differences in the progression of HIV infection in hemophiliacs.

DETAILED DESCRIPTION:
BACKGROUND:

In the late 1980s, hemophiliacs were transfused with a variety of blood products, including large amounts of cryoprecipitate. In comparison to other cohorts, hemophiliacs are CMV(-), resulting in a comparison group for the study of this virus as a potential cofactor. In contrast, non A, non-B hepatitis is common in comparison to other cohorts, and preliminary data prior to 1990 suggested that this chronic disease predisposes to more rapid progression of HIV infection.

DESIGN NARRATIVE:

Disease-free survival rates were determined in HIV-infected hemophiliacs. The effects of co-factors such as intensive transfusion, concomitant cytomegalovirus or chronic NANB hepatitis infection were ascertained. Host-virus interaction was assessed through the use of plasma cultures, specific antibody titers, and markers of immune changes detected by flow cytometry and immune function assays. The immunology of asymptomatic stable infection was investigated. The safety of volunteer donor blood products was determined in seronegative patients exposed to over 50,000 donors yearly and the risk of sexual transmission of HIV to spouses of seropositive patients was monitored.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-07 (Actual); Primary Completion 1995-03 (Actual); Study Completion 1995-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Gjerset — Bloodworks